CLINICAL TRIAL: NCT03329287
Title: Efficacy, Prediction and Methodological Evaluation of Simplified Cognitive Behavioral Therapy for Generalized Anxiety Disorder and Depression: a Multicenter, Randomized, Controlled Study
Brief Title: Simplified Cognitive Behavioral Therapy for Generalized Anxiety Disorder and Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: Changhai Hospital (Other); Shanghai 10th People's Hospital (Other); Tongji Hospital (Other); Fudan University (Other); Second Hospital of Shanxi Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15411950201
Record Dates: First submitted 2017-10-26; First posted 2017-11-01 (Actual); Last update posted 2017-11-01 (Actual); Status verified 2017-07

CONDITIONS: Generalized Anxiety Disorder; Major Depressive Disorder
Keywords: Simplified Cognitive Behavioral Therapy (SCBT); Generalized Anxiety Disorder; Depression; Operating manual; Efficacy
MeSH Terms: conditions — Generalized Anxiety Disorder; Depressive Disorder, Major; Depression | interventions — Serotonin and Noradrenaline Reuptake Inhibitors

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SCBT + Drug (Experimental): Participants receive SCBT at a frequency of twice a week in the first 4 weeks, and once a week in the following 4 weeks. They also take SSRIs and/or SNRIs through the trial at a recommended dosage.
  Interventions: Behavioral: SCBT; Drug: SSRIs and/or SNRIs
- Psychological Placebo + Drug (Active Comparator): Participants receive supportive and relaxation therapy at a frequency of twice a week in the first 4 weeks, and once a week in the following 4 weeks. They also take SSRIs and/or SNRIs through the trial at a recommended dosage.
  Interventions: Drug: SSRIs and/or SNRIs; Behavioral: Psychological Placebo
- Drug (Active Comparator): Participants only take SSRIs and/or SNRIs through the trial at a recommended dosage.
  Interventions: Drug: SSRIs and/or SNRIs

INTERVENTIONS:
Behavioral: SCBT — SCBT, one hour per session.
  Arms: SCBT + Drug
Drug: SSRIs and/or SNRIs — SSRIs and/or SNRIs at a recommended dosage.
Behavioral: Psychological Placebo — Supportive and relaxation therapy, one our per session.
  Arms: Psychological Placebo + Drug

SUMMARY:
This trial attempts to evaluate the treatment efficacy of Simplified Cognitive Behavioral Therapy (SCBT) and its safety among schizophrenia patients. Half of participants will be randomized to accept SCBT.

DETAILED DESCRIPTION:
The investigators have developed a simplified but standardized set of cognitive behavioral treatment (including the therapist's manual and patient self-help manual) for the patients of generalized anxiety disorder and depression, known as Simplified Cognitive Behavioral Therapy (SCBT). SCBT is the main psychological intervention of this study. The aim of this study is to verify its efficacy and applicability using a multi-center, randomized, placebo controlled and single-blind design, and to optimize the treatment program. The investigators hypothesize that SCBT is effective in patients with depression or anxiety, and the manual is easily-operated for the therapists.

ELIGIBILITY:
Inclusion Criteria:

* 1. Adults aged 18-60 years old, male and female; 2. With primary school or above education levels; 3. Without vision, hearing or communication difficulties; 4. DSM-V diagnosis of generalized anxiety disorder and/or major depressive disorder; 5. HAMA-14 score greater than or equal to 14 points, less than 29 pionts; HAMD-17 score greater than or equal to 7 points, less than 24 points; 6. GAD-7 score greater than or equal to 5 points; PHQ-9 score greater than or equal to 5 points; 7. In the last 2 months, did not accept other forms of psychological treatment, or treatment is ineffective; 8. Voluntarily participate in and sign informed consent.

Exclusion Criteria:

1. Suffering from serious physical illness;
2. Having self-injurious behavior, suicidal tendencies;
3. Having bipolar disorder;
4. Having psychotic symptoms;
5. Having obsessive-compulsive disorder, post-traumatic stress disorder;
6. Pregnant women or lactating women.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-03-30 (Estimated); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
changes of The Hamilton Depression Scale (HAMD-17) | At baseline, 2-week, 4-week, 6-week, 8-week, 12-week, 20-week, 32-week and 56-week.
  Scale total range is 52. Lower score represents a better outcome.
changes of The Hamilton Anxiety Scale (HAMA-14) | At baseline, 2-week, 4-week, 6-week, 8-week, 12-week, 20-week, 32-week and 56-week.
  Scale total range is 56. Lower score represents a better outcome.

SECONDARY OUTCOMES:
changes of The Patient Health Questionnaire (PHQ-9) | At baseline, 2-week, 4-week, 6-week, 8-week, 12-week, 20-week, 32-week and 56-week.
  Scale total range is 27. Lower score represents a better outcome.
changes of The GAD-7 | At baseline, 2-week, 4-week, 6-week, 8-week, 12-week, 20-week, 32-week and 56-week.
  Scale total range is 21. Lower score represents a better outcome.
changes of The Mos 36-item Short Form Health Survey (SF-36) | At baseline, 4-week, 8-week, 12-week, 20-week, 32-week and 56-week.
  It has nine dimensions, each dimension has an independent fractional formula.
changes of Treatment Emergent Symptom Scale (TESS) | At baseline, 2-week, 4-week, 6-week, 8-week, 12-week, 20-week, 32-week and 56-week.
  Evaluation of side effects caused by various psychotropic drugs.
changes of Clinical Global Impression (CGI) | At baseline, 2-week, 4-week, 6-week, 8-week, 12-week, 20-week, 32-week and 56-week.
  Evaluation of clinical efficacy. Lower score represents a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Chunbo Li, PHD, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD data